OnabotA X 2042-201-008 – Statistical Analysis Plan Version 2.0 – 12 December 2022

## Statistical Analysis Plan for Study 2042-201-008

A Multicenter, Double-Blind, Randomized,
Placebo-Controlled Parallel-Group Phase 2 Study
Evaluating the Safety and Efficacy of
OnabotulinumtoxinA X for the Treatment of
Moderate to Severe Glabellar Lines

Date: 12 December 2022

Version 2.0

# **Table of Contents**

| 1.0 | Introduction | 5 |
|---|---|---|
| 2.0 | Study Design and Objectives | 5 |
| 2.1 | Objectives, Hypotheses and Estimands | 5 |
| 2.2 | Study Design Overview | 6 |
| 2.3 | Treatment Assignment and Blinding | 7 |
| 2.4 | Sample Size Determination | 7 |
| 3.0 | Endpoints | 8 |
| 3.1 | Primary Endpoint(s) | 8 |
| 3.2 | Secondary Endpoint(s) | 8 |
| 3.3 | Other Efficacy Endpoint(s) | 8 |
| 3.4 | Safety Endpoint(s) | 10 |
| 3.5 | Additional Endpoint(s) | 11 |
| 4.0 | Analysis Populations | 11 |
| 5.0 | Subject Disposition | 12 |
| 6.0 | Study Drug Duration and Compliance | 12 |
| 7.0 | Demographics, Baseline Characteristics, Medical History, and Prior/Concomitant Medications | 12 |
| 7.1 | Demographics and Baseline Characteristics | |
| 7.2 | Medical History | 13 |
| 7.3 | Prior and Concomitant Medications | |
| 7.4 | Concurrent Procedure | 14 |
| 8.0 | Handling of Potential Intercurrent Events for the | 1.4 |
| 9.0 | Primary and Key Secondary Endpoints<br>Efficacy Analyses | |
| 9. <b>0</b><br>9.1 | General Considerations | |
| 9.1<br>9.2 | | |
| - | Handling of Missing Data | |
| 9.3 | Primary Efficacy Endpoint(s) and Analyses | |
| 9.3.1 | Primary Efficacy Endpoint(s) | |
| 9.3.2 | Main Analysis of Primary Efficacy Endpoint(s) | 17 |
| 9.3.3 | Sensitivity and Supplementary Analyses of the Primary Efficacy Endpoint(s) | 18 |

# OnabotA X 2042-201-008 – Statistical Analysis Plan Version 2.0 – 12 December 2022

| 9.4 | Secondary Efficacy Endpoints and Analyses | 18 |
|---|---|---|
| 9.4.1 | Key Secondary Efficacy Endpoints | |
| 9.4.2 | Main Analyses of Key Secondary Efficacy Endpoints | 19 |
| 9.4.3 | Sensitivity and Supplementary Analyses for Key Secondary Efficacy Endpoints | |
| 9.4.4 | Supportive Secondary Efficacy Endpoints and Analyses | 21 |
| 9.5 | Additional Efficacy Analyses | 21 |
| 9.6 | Efficacy Subgroup Analyses | 23 |
| 10.0 | Safety Analyses | 23 |
| 10.1 | General Considerations | 23 |
| 10.2 | Adverse Events | 23 |
| 10.2.1 | Treatment-Emergent Adverse Events | 23 |
| 10.2.2 | Adverse Event Overview | 24 |
| 10.2.3 | Treatment-Emergent Adverse Events by SOC and/or PT | 24 |
| 10.2.4 | SAEs (Including Deaths) and Adverse Events Leading to Study<br>Drug Discontinuation | 25 |
| 10.2.5 | Potential Distant Spread of Toxin Adverse Events | 25 |
| 10.3 | Analysis of Laboratory Data | 25 |
| 10.4 | Analysis of Vital Signs | 26 |
| 10.5 | Safety Subgroup Analyses | 27 |
| 10.6 | Other Safety Analyses | 27 |
| 11.0 | Other Analyses | 28 |
| 12.0 | Interim Analyses | 28 |
| 12.1 | Data Monitoring Committee | 29 |
| 13.0 | Overall Type-I Error Control | 29 |
| 14.0 | Version History | 30 |
| 15.0 | References | 30 |
| List of Table 1. | | |
| rable 1. | Summary of the Estimand Attributes of the Primary Efficacy Endpoint | 17 |



OnabotA X
2042-201-008 – Statistical Analysis Plan
Version 2.0 – 12 December 2022

| Table 2. | Summary of the Estimand Attributes of the Secondary Efficacy | |
|---|---|---|
| | Endpoints | 20 |
| Table 3. | SAP Version History Summary | 30 |
| List of Fig | ures | |
| 3 | | |
| Figure 1. | Study Schematic | 7 |
| List of App | pendices | |
| Appendix A. | Protocol Deviations | 31 |
| Appendix B. | Definition of Possible Distant Spread of Toxin | 32 |
| Appendix C. | Potentially Clinically Important Criteria for Safety Endpoints | 33 |



#### 1.0 Introduction

This Statistical Analysis Plan (SAP) describes the statistical analyses for OnabotA X Study 2042-201-008 Glabellar Lines: OnabotulinumtoxinA X in the Treatment of Moderate to Severe Glabellar Lines.

Study 2042-201-008 examines the safety and efficacy of OnabotA X in subjects with moderate to severe glabellar lines.

The SAP will not be updated in case of administrative changes or amendments to the protocol unless the changes impact the analysis.

Unless noted otherwise, all analyses will be performed using SAS Version 9.4 (SAS Institute Inc., Cary, NC 27513) or later under the Linux operating system.

#### 2.0 Study Design and Objectives

#### 2.1 Objectives, Hypotheses and Estimands

The primary objectives of the study are to compare the efficacy of OnabotA X and placebo and to evaluate the safety of OnabotA X in subjects with moderate to severe GL.

The null and alternate hypotheses are the following:

 $H_0$ :  $P_T = P_P$  (The treatment response probability between each OnabotA X treatment group and the placebo group is equal)

 $H_A$ :  $P_T \neq P_P$  (The treatment response probability between each OnabotA X treatment group and the placebo group is not equal)

Estimand attributes of the primary efficacy endpoint are detailed in Table 1 (see Section 9.3.2). In addition, the attribute of treatment is a single dose of active treatment or placebo.

Differences in proportion of subjects who would achieve ≥ 1-grade improvement from baseline on the investigator-rated AGLSS at maximum contraction at Day 30 had they not



missed AGLSS assessments, for each active treatment group (OnabotA X ) in comparison with placebo in the ITT population.

Any missing assessments will be assumed to be missing at random and imputed using multiple imputation. Statistical significance of the difference will be tested using Cochran-Mantel-Haenszel (CMH) test stratified by baseline investigator-rated AGLSS at maximum contraction.



The clinical hypothesis is that OnabotA X has an acceptable safety profile when administered to the corrugator and procerus muscles in subjects with moderate to severe GL.

No estimand is defined for the safety evaluations.

## 2.2 Study Design Overview

The schematic of the study is shown in Figure 1.

Figure 1. Study Schematic



#### 2.3 Treatment Assignment and Blinding

Subjects will be randomized in a 2:2:2:1 ratio to receive OnabotA X placebo or placebo or Randomization will be stratified at each investigator site by baseline investigator-rated AGLSS at maximum contraction, using central by block stratified randomization. The same block will not be shared across investigative sites or by baseline GL severity assessment. AbbVie will provide instructions for preparations and treatment administration separately, in the pharmacy manual.

# 2.4 Sample Size Determination

| The sample size was chosen empirically. |
|-----------------------------------------|









# 3.4 Safety Endpoint(s)

The safety endpoints for this study include:

- Adverse Events
- Abbreviated Physical Examination (general appearance, head, ears, eyes, nose, throat, and neck)



| | Clinical Laboratory Test |
|---|---|
| | Vital Sign Measurements |
| | • Electrocardiogram |
| | Neurologic Assessment |
| 3.5 | Additional Endpoint(s) |
| 4.0 | Analysis Populations |
| The fol | llowing population sets will be used for the analyses. |
| | tent to Treat (ITT) Population includes all randomized subjects. The ITT |
| Popula | tion will be used for all efficacy analyses. |
| | fety Analysis Set consists of all subjects who received at least 1 dose of study drug. fety analyses will be based on the safety population. |

# 5.0 Subject Disposition

The total number of subjects who were screened, enrolled, and treated will be summarized. Reasons for exclusion, including screen failure, will be summarized.



For end of study participation, the number and percentage of subjects who completed the protocol defined follow-up period (or did not with associated reasons) will be summarized overall and by treatment group.

# 6.0 Study Drug Duration and Compliance

Duration of exposure will be summarized with descriptive statistics (mean and standard deviation, median, Q1, Q3, minimum, and maximum). The number of subjects exposed for specific period of time

will also

be summarized. Duration of exposure will be calculated as data of study exit minus data.

be summarized. Duration of exposure will be calculated as date of study exit minus date of study drug administration +1.

# 7.0 Demographics, Baseline Characteristics, Medical History, and Prior/Concomitant Medications

Demographics, baseline characteristics, medical history, prior and concomitant medications, and concurrent procedure will be summarized overall and by treatment group for the ITT Population.



| 7.1 | Demographics and Baseline Characteristics |
|---|---|
| | mographic variables include age. Categorical demographic variables unicity, race, age group |
| type, investiga | cteristics include weight, height, body mass index (BMI), Fitzpatrick skin tor-rated and subject-rated AGLSS severity at maximum contraction and a facial Line Satisfaction Questionnaire (FLSQ <sup>©</sup> ) impact domain score, |
| 7.2 | Medical History |
| Medical history (MedDRA). | y data will be coded using the Medical Dictionary for Regulatory Activities |
| 7.3 | Prior and Concomitant Medications |
| Prior and conc | omitant medications will be summarized by generic name. |



number and percentage of subjects taking medications will be summarized by generic drug name based on the World Health Organization (WHO) Drug Dictionary for both prior and concomitant medications. 7.4 **Concurrent Procedure** All procedures undergone on or after Study Day 1 visit through the exit visit will be considered concurrent procedures. Concurrent procedure will be summarized by MedDRA high level term and preferred term. **Handling of Potential Intercurrent Events for the** 8.0 **Primary and Key Secondary Endpoints** The primary endpoint and secondary endpoints will be analyzed based on the ITT population,



• Subjects who are missing data for any other reason for the endpoint will count as though they hypothetically continued in the study.

#### 9.0 Efficacy Analyses

#### 9.1 General Considerations



Unless otherwise specified, any subject who is randomized based on a wrong stratum will be analyzed according to the actual stratum the subject belongs to.

"Baseline" refers to the last non-missing observation before the first administration of study drug or randomization if no study drug is given.

#### 9.2 Handling of Missing Data

Missing data will be imputed using multiple imputation (MI) method for the primary and secondary endpoints.





Each of the 5 imputation data sets will be analyzed individually, then combined to generate the final inferences as described in Section 9.3.2.

#### 9.3 Primary Efficacy Endpoint(s) and Analyses

#### 9.3.1 Primary Efficacy Endpoint(s)

The primary efficacy endpoint is achievement of  $\geq$  1-grade improvement from baseline on the investigator-based AGLSS at maximum contraction at Day 30.

#### 9.3.2 Main Analysis of Primary Efficacy Endpoint(s)

The attributes of the estimands corresponding to the primary efficacy endpoint are summarized in Table 1.

Table 1. Summary of the Estimand Attributes of the Primary Efficacy Endpoint

| | Attributes of the Estimand | | | | |
|---|---|---|---|---|---|
| Estimand<br>Label | Treatment | Endpoint | Population | Handling of Intercurrent Events | Statistical<br>Summary |
| Hypothetical estimand for primary endpoint | OnabotA X or placebo | Achievement of ≥ 1-grade improvement from baseline on the AGLSS according to investigator assessments at maximum contraction at Day 30 | ITT (All randomized) | Subjects who discontinue study prior to Day 30 assessments, or who do not have AGLSS assessments will be included in the analysis as a hypothetical scenario in which they had not missed the AGLSS assessments | Difference in response proportions between each active treatment group and placebo, after MI using CMH test stratified by baseline investigatorrated AGLSS at maximum contraction |

AGLSS = Allergan Glabellar Line Severity Scale; CMH = Cochran-Mantel-Haenszel; ITT = intent-to-treat; MI = multiple imputation; OnabotA X = onabotulinumtoxinA X

The evaluation of the equality of the proportions of responders will be based on Cochran-Mantel-Haenszel (CMH) test stratified by baseline investigator-rated AGLSS at maximum contraction. Wald confidence intervals for proportions of responders and difference in the proportion of responders will be presented. The Breslow-Day homogeneity of the odds-



ratio test will be performed to test the treatment-by-investigator-rated baseline GL severity at maximum contraction interaction.

To obtain pooled CMH p-value, the Wilson-Hilferty transformation will be used.<sup>1,2</sup>

# 9.3.3 Sensitivity and Supplementary Analyses of the Primary Efficacy Endpoint(s)

A sensitivity analysis will be performed for the primary efficacy variable using observed data.

#### 9.4 Secondary Efficacy Endpoints and Analyses

#### 9.4.1 Key Secondary Efficacy Endpoints

The key secondary endpoints, which utilize both the AGLSS and FLSQ, include:

- Achievement of None or Mild on the investigator-rated AGLSS assessments at maximum contraction at Day 30;
- Responses of Very satisfied or Mostly satisfied on satisfaction with treatment per the FLSQ follow-up version Item 5 at Day 60;
- Achievement of ≥ 14-point psychosocial impact improvement from baseline at Day 30 per the FLSQ Impact domain, among subjects with baseline scores ≥ 14 points



# 9.4.2 Main Analyses of Key Secondary Efficacy Endpoints

The attributes of the estimands corresponding to the secondary efficacy endpoints are summarized in Table 2.



Table 2. Summary of the Estimand Attributes of the Secondary Efficacy Endpoints

| | Attributes of the Estimand | | | | |
|---|---|---|---|---|---|
| Estimand<br>Label | Treatment | Endpoint | Population | Handling of<br>Intercurrent Events | Statistical<br>Summary |
| Hypothetical estimand for secondary endpoint | OnabotA X or placebo | Achievement of<br>None or Mild on<br>the investigator-<br>rated AGLSS<br>assessments at<br>maximum<br>contraction at<br>Day 30 | ITT (All randomized) | Subjects who discontinue study prior to Day 30 assessments, or who do not have AGLSS assessments will be included in the analysis as a hypothetical scenario in which they had not missed the AGLSS assessments | Difference in response proportions between each active treatment group and placebo, after MI using CMH test stratified by baseline investigator- rated AGLSS at maximum contraction |
| | | Responses of<br>Very satisfied or<br>Mostly satisfied<br>on satisfaction<br>with treatment<br>per the FLSQ<br>follow-up<br>version Item 5 at<br>Day 60 | Subjection Date of the Date of | Subjects who discontinue study prior to Day 60 assessments, or who do not have FLSQ assessments will be included in the analysis as a hypothetical scenario in which they had not missed the FLSQ assessments | |
| | | Achievement of ≥ 14-point psychosocial impact improvement from baseline at Day 30 per the FLSQ Impact domain, among subjects with baseline scores ≥ 14 points | _ | Subjects who discontinue study prior to Day 30 assessments, or who do not have FLSQ assessments will be included in the analysis as a hypothetical scenario in which they had not missed the FLSQ assessments | _ |

 $AGLSS = Allergan \ Glabellar \ Line \ Severity \ Scale; CMH = Cochran-Mantel-Haenszel; \ ITT = intent-to-treat; \\ MI = multiple \ imputation; \ OnabotA \ X = onabotulinum toxinA \ X$ 



The key secondary efficacy endpoints are to be analyzed similarly to the primary endpoint using multiple imputation, as specified in Section 9.2.

9.4.3 Sensitivity and Supplementary Analyses for Key Secondary Efficacy Endpoints

Not applicable.

9.4.4 Supportive Secondary Efficacy Endpoints and Analyses

Not applicable.

9.5 Additional Efficacy Analyses







| 9.6 | Efficacy Subgroup Analyses |
|---|---|
| Not applicable. | |
| 10.0 | Safety Analyses |
| 10.1 | General Considerations |
| • | e summarized for the Safety Analysis Set. For the safety analyses, narized based on the treatment actually received. |
| 10.2 | Adverse Events |
| using primary Me | Adverse events (AEs) will be summarized overall and by treatment group and presented using primary MedDRA System Organ Classes (SOCs) and preferred terms (PTs) according to the version of the MedDRA coding dictionary used for the study at the time |
| of database lock. | |
| 10.2.1 | Treatment-Emergent Adverse Events |
| | All treatment-emergent AEs will be summarized |
| overall, as well as | s by primary MedDRA SOC and Preferred Term. |



#### 10.2.2 Adverse Event Overview

An overview of AEs will be presented consisting of the number and percentage of subjects experiencing at least one event for each of the following AE categories:

- Any treatment-emergent AE
- Any treatment-emergent AE related to study treatment according to the investigator



- Any PDSOT TEAEs
- All deaths

#### 10.2.3 Treatment-Emergent Adverse Events by SOC and/or PT

Treatment-emergent AEs will be summarized by system organ class (SOC) and PT; by maximum severity and SOC and PT; and by subject number and SOC and PT.

| 10.2.4 | SAEs (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation |
|---|---|
| SAEs (includ | ding deaths) will be summarized by SOC and PT and in listing format. |
| 10.2.5 | Potential Distant Spread of Toxin Adverse Events |
| To assess PI | OSOT, MedDRA preferred terms that may be associated with botulinum toxing |
| | been identified (Appendix B). |
| 10.3 | Analysis of Laboratory Data |
| | The clinical |
| _ | sts defined in the protocol operations manual (e.g., hematology, clinical nd urinalysis) will be summarized by treatment group. |

| 10.4 | Analysis of Vital Signs |
|---|---|
| | rements of systolic and diastolic blood pressure, pulse rate, respiratory emperature will be summarized by treatment group. |

| | <del>-</del> |
|------------------------|--------------------------|
| 10.5 | Safety Subgroup Analyses |
| Not applicable. | |
| 10.6 | Other Safety Analyses |
| 10.6 Electrocardiogran | |

| Neurologic A | Assessment: |
|---|---|
| 1 tearorogie 1 | <u>kobedsirient.</u> |
| 11.0 | Other Analyses |
| <u>Immunogeni</u> | city: Blood samples for immunogenicity testing will be collected from all |
| subjects | |
| Hypersensiti | vity: Blood samples to be collected within 2 hours of suspected anaphylaxis |
| or systemic h | hypersensitivity reaction. |
| 12.0 | Interim Analyses |
| A | |
| An interim a | nalysis is planned to occur If a dose recommendation cannot be made at this |
| point, then a | second interim analysis will be performed |
| point, then to | The interim analyses will be comparative and will be |
| unblinded to | a group of AbbVie personnel who are not directly involved in ongoing day- |
| to-day study | conduct. |
| | Further details are provided in DMC Charter. |
| The primary | and secondary efficacy analyses will be performed for each interim analysis, |
| | mmaries of all safety variables. |

# 12.1 Data Monitoring Committee

| An independ | lent DMC will be instituted to review interim safety and efficacy data to |
|---|---|
| provide a do | se recommendation for Phase 3. A DMC Charter will be finalized prior to |
| study start. | |
| 13.0 | Overall Type-I Error Control |
| Analyses wi | Il be conducted using a gated hierarchical testing procedure to preserve a |
| _ | Type I error rate of $\alpha$ =0.05 for each OnabotA X group compared to placebo, |
| separately. | |
| 1 7 | |

# 14.0 Version History

**Table 3. SAP Version History Summary** 

| Version | Date of Approval | Summary |
|---|---|---|
| 1.0 | 19 August 2021 | Initial version |
| 2.0 | | Section 2.1, added details for estimand |
| | | Section 4.0, changed the safety analysis set to be analyzed per<br>randomization due to the difficulty of determine the actual<br>treatment |
| | | Section 8.0, added details for handling potential intercurrent events |
| | | Section 9.3.2 Table 1, updated column 'Handling of Intercurrent Events' |
| | | Section 9.4.2 added Table 2, the Summary of the Estimand Attributes of the Secondary Efficacy Endpoints |
| | | Updated Table B-1 MedDRA preferred terms evaluated for PDSOT, removed the term "Extraocular muscles paresis", added the term "Opthalmoplegia" |
| | | Updated Table C-1 Criteria for Potentially Clinically Important<br>Clinical Laboratory Values: updated the value corresponding to<br>Cholesterol, Glucose, and Triglycerides. Changed "Inorganic<br>phosphorus" to "Phosphate" |

# 15.0 References

- 1. EB W, MM H. The distribution of chi-square. Proc Natl Acad Sci U S A. 1931;17(12):684-8.
- 2. O'Kelly M, Ratitch B. Clinical trials with missing data: a guide for practitioners. First ed: John Wiley & Sons, Ltd; 2014.



#### **Appendix A.** Protocol Deviations

The number and percentage of unique subjects reporting significant protocol deviations will be summarized in total and by treatment group for all randomized or treated subjects. The number and percentage of unique subjects with protocol deviation categories below will also be summarized in total and by treatment group.

- Subject entered into the study even though s/he did not satisfy entry criteria.
- Subject received wrong treatment or incorrect dose of study.
- Subject took prohibited concomitant medication or concurrent procedure.



## Appendix B. Definition of Possible Distant Spread of Toxin

#### Table B-1. MedDRA Preferred Terms Evaluated for PDSOT

| Accommodation disorder | Hyporeflexia |
|--------------------------------|------------------------------|
| Aspiration | Hypotonia |
| Bell's Palsy | Ileus paralytic |
| Botulism | Muscular weakness |
| Bradycardia | Opthalmoplegia |
| Bulbar palsy | Paralysis |
| Constipation | Paresis cranial nerve |
| Cranial nerve palsies multiple | Pelvic floor muscle weakness |
| Cranial nerve paralysis | Peripheral nerve palsy |
| Diaphragmatic paralysis | Peripheral paralysis |
| Diplopia | Pneumonia aspiration |
| Dry mouth | Pupillary reflex impaired |
| Dysarthria | Respiratory arrest |
| Dysphagia | Respiratory depression |
| Dysphonia | Respiratory failure |
| Dyspnoea | Speech disorder |
| Eyelid function disorder | Urinary retention |
| Eyelid ptosis | Vision blurred |
| Facial paralysis | Vocal cord paralysis |
| Facial paresis | Vocal cord paresis |

Note: Table is based on MedDRA 25.0; the actual list used for analysis will be based on the MedDRA version in use at the time of database lock.







